CLINICAL TRIAL: NCT05667675
Title: Targeting Child Mental Health and Household Poverty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imaan Bayoumi (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor-Investigator, Imaan Bayoumi, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEAMO IF Bayoumi
Record Dates: First submitted 2022-12-10; First posted 2022-12-28 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2023-11

CONDITIONS: Poverty; Child Health; Behavior Problem
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: A pragmatic, 1:1 allocation, parallel-group superiority pilot randomized controlled trial will be conducted.
Who Masked: Investigator, Outcomes Assessor
Masking Description: It will not be possible to blind participants to their group allocation. However, study information materials and the consent form will indicate that after consenting they will be randomly allocated to one of two approaches to providing support, without a detailed description of the interventions. This approach will provide some degree of blinding of participants. Additionally, RAs conducting outcomes assessment visits, the biostatistician and investigators will remain blind to each child's group allocation. Blinding will be achieved by having the group allocation coded as A and B in the database; group allocation will be concealed until the final data analysis is performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community Support Worker (Experimental): Participants in the intervention group will have a structured review of their financially related needs and resources with a trained CSW, who will have a thorough understanding of potential income supports and community support agencies. The CSW will use a structured approach to identify financial needs and benefits for which the family is eligible The CSW will work intensively with families in the intervention arm to identify and meet their goals. They will conduct weekly meetings to complete forms, and provide advocacy (in person and by telephone) as needed up to six meetings as needed for system navigation.
  Interventions: Behavioral: Community Support Worker
- Control (Active Comparator): There is no clear standard of care and potential for practice variation in clinician responses to identified social need. For this proposal, participants in the comparator group will receive Usual care, defined as: Participants in both groups will receive a written summary of available resources.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Community Support Worker — Participants in the intervention group will have a structured review of their financially related needs and resources with a trained CSW, who will have a thorough understanding of potential income supports and community support agencies. The CSW will use a structured approach to identify financial needs and benefits for which the family is eligible The CSW will work intensively with families in the intervention arm to identify and meet their goals. They will conduct weekly meetings to complete forms, and provide advocacy (in person and by telephone) as needed up to six meetings as needed for system navigation.
  Arms: Community Support Worker
Behavioral: Control — There is no clear standard of care and potential for practice variation in clinician responses to identified social need. For this proposal, participants in the comparator group will receive Usual care, defined as: Participants in both groups will receive a written summary of available resources.
  Arms: Control

SUMMARY:
Living in poverty has long-lasting negative effects on children's mental health and on their mental health in adulthood. Child poverty is very common, affecting 17% of Canadian children. Many low income families may not be getting all the social benefits they are entitled to receive. Increasingly, there are calls for primary care providers to ask all patients about poverty and to intervene if poverty is identified. However, it is not known if an intervention can improve children's health. This study will test the effect of having a Community Support Worker work with families of children age 2-5 years during a primary care visit to identify unmet financially related social needs (like food, housing or energy insecurity) and help families navigate the social service system. The Community Support Worker will help families complete income tax, apply for benefits and community supports to which they are entitled. The investigators will study the effect on child emotional and behavioural health, parent stress and depression and family income. Results from this study will help health care providers and policy makers understand whether this is an effective way to integrate the health and social service systems to improve child and parent health.

DETAILED DESCRIPTION:
Background: Child poverty remains a prevalent problem in Canada, affecting 17% of Canadian children. There are profound negative impacts on child health related to poverty, particularly when the exposure is prolonged or occurs in early childhood, affecting mental health (higher prevalence of depression, conduct disorders and ADHD) and school readiness. Socio-economic health disparities are estimated to cost the health care system $6.2 billion annually. Moreover, investments in early childhood have an estimated annual return of investment of 7-10%.

Emotional and behavioural problems, including depression, anxiety, conduct and hyperactivity problems) serious enough to impair daily function occur in 14-26% of preschool children, with increased risk in low income families and those with lower parental education. Furthermore, vulnerability in emotional and behavioural domains in Kindergarten is associated with poor future academic performance and is more prevalent in low income families. Poor mental health trajectories in preschool age children are associated with high family stress and maternal depression. In turn, reduced family stress is associated with fewer child behaviour problems. Additionally, chronic exposure to poverty has been associated with poor mental health along a gradient, in which those most affected were always poor, followed by those experiencing intermittent poverty and finally, those least affected were never poor.

An estimated 40-60% of preschool children with significant emotional and behavioural symptoms will continue to experience problems 10 years later and are at increased risk for mental health problems in adulthood. A growing body of scientific evidence demonstrates the mechanisms by which social and environmental early life exposure directly influences the architecture of the young developing brain. Both the Canadian Paediatric Society and the American Academy of Pediatrics take the position that "adult diseases should be viewed as developmental disorders beginning early in life and that persistent health disparities associated with poverty, discrimination and maltreatment can be reduced by the alleviation of toxic stress in childhood". Poverty has been associated with demonstrated changes in brain architecture, affecting the temporal lobe, amygdala, hippocampus and prefrontal cortex, areas of the brain critical to decision making, emotional regulation, mood and impulse control, language development and memory. Such permanent early changes in brain development establish a poor foundation for future mental health and learning and help to explain persistent health, educational and social disparities. Given the long-term impact of childhood poverty on overall health, effective interventions have the potential to translate into improved health outcomes and significant healthcare savings.

Community Support Workers: Community Support Workers (CSW) provide health education, anticipatory guidance, supported attendance at medical appointments and adherence to medically recommended care to families. These visits have been shown to improve immunization rates, and access to dental care. However, their role in addressing poverty and other unmet social needs and child behavioural health has not been studied. The CSW role has been implemented in the SELHIN in several primary care settings with the goal of addressing unmet social needs for high need patients. CSWs have a thorough understanding of available income supports and community support agencies and review social needs, such as food, housing and energy insecurity. They help patients access social benefits for which they are eligible, including ensuring up-to-date completion of income tax returns, application for disability benefits, benefits such as the Special Diet allowance, and other programs. The tax system is the principal policy mechanism to provide critically needed social benefits to Canadians, however many eligible Canadians lack the awareness, knowledge and confidence to access all benefits they are entitled to receive. Many low income Canadians, particularly those facing additional barriers such as women living with their children in shelters, Indigenous people and young parents, have disproportionately lower tax filing rates and are therefore not benefiting from many government social supports. The impact of the Canada Child Benefit, established in 2016 is still not known; however,it is likely that many eligible families have not applied. The impact of this integrated income support role in primary care on child and parent health is not known. Addressing this knowledge gap will inform policy changes, potentially encouraging scaling up the CSW role to additional primary care models, including team-based, sole proprietor family medicine, pediatrics and nurse practitioner led clinics.

This project builds on a previously funded SEAMO IF project, 'Implementation of a clinical poverty intervention tool --Phase 1: Process evaluation', which determined that poverty screening by physicians was seen as important by clinicians and highly acceptable to patients. Clinicians found universal screening to be difficult, in part because they were not confident in their ability to address identified needs. This project builds on these findings by embedding and evaluating an intervention, which will establish the health outcomes associated with a structured poverty intervention.

Significance and innovation: A recent systematic review summarized the literature on health care interventions to address unmet social needs in the U.S. A single study examining child health outcomes associated with an intervention targeting income security, found fewer social needs and improved caregiver reported overallchild health.26 To date, the health outcomes for children or parents associated with poverty screening in Canadian health care settings, in the context of universally available healthcare have not been evaluated. There is consensus on the need to address social determinants to improve health and reduce health system costs, but little is known about effective interventions. Specifically, it is unclear whether structured review of financially-related social needs and social system navigation for low income families can improve child emotional and behavioural health and parent mental health outcomes.

Objective: To execute an internal pilot study, in preparation for a multi-site full trial to determine if structured review of financially-related social needs and social system navigation for low income families can improve child emotional and behavioural health and reduce parent stress and depression.

Rationale: Health care providers increasingly endorse the importance of social needs and good health but report low confidence in their ability to meet their patients' unmet social needs. The College of Family Physicians of Canada (CFPC) recommends screening patients using the single question "Do you ever have difficulty making ends meet at the end of the month?" However, neither screening nor intervention tools are routinely used in primary practice and to date, the impact of poverty screening on health outcomes has not been evaluated in Canada.

Specific Hypotheses of the Internal Pilot:

1. Randomization rate: there is a reasonably high probability that at least 50% of approached parents will agree to randomization.
2. Retention and completion rate: there is a reasonably high probability that at least 80% of participants will complete the trial.
3. Feasibility of primary and secondary outcomes: there is a reasonably high probability that at least 80% of participants will complete the primary and secondary outcomes.
4. Sample size estimates: The standard deviation for the primary outcome used to determine the sample size for the full trial is no less than 10% lower than the one observed in the pilot.

ELIGIBILITY:
Inclusion Criteria:

* Children age 2-5y attending a routinely scheduled visit with their primary care provider. - - Parents respond affirmatively to the question "Do you ever have difficulty making ends meet at the end of the month?"
* Informed parental consent. Only one child will be enrolled per family. For families with more than one child, we will enroll the youngest eligible child.

Exclusion Criteria:

* Child born prematurely (gestational age less than 32 weeks)
* birthweight less than 2500g
* Parent unable to communicate in English.
* Parents without legal status in Canada.
* Families already receiving support with system navigation, such as from a social worker or public health nurse.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire, Total Difficulties Score | 6 months after enrollment.
  A validated 25 item mental health questionnaire for children 2-17 years old on 5 domains (emotional problems, conduct problems, hyperactivity/inattention, peer problems and a prosocial scale). The first 4 scales are combined to give a Total Difficulties Score. Items in the first four scales are assigned a score of 0-2 (0 indicates 'Not True', 1 indicates 'Somewhat True' and 2 indicates 'Certainly True'). Reverse scoring is used for the Prosocial scale. Subscale totals range from 0-10 and the Total Difficulties Score can range from 0-40. Higher scores reflect greater difficulties for the Difficulties scores, and greater prosocial behaviour for the Prosocial score.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire, Total Difficulties Score | 12 months after enrollment
  A validated 25 item mental health questionnaire for children 2-17 years old on 5 domains (emotional problems, conduct problems, hyperactivity/inattention, peer problems and a prosocial scale). The first 4 scales are combined to give a Total Difficulties Score. Items in the first four scales are assigned a score of 0-2 (0 indicates 'Not True', 1 indicates 'Somewhat True' and 2 indicates 'Certainly True'). Reverse scoring is used for the Prosocial scale. Subscale totals range from 0-10 and the Total Difficulties Score can range from 0-40. Higher scores reflect greater difficulties for the Difficulties scores, and greater prosocial behaviour for the Prosocial score.

OTHER OUTCOMES:
Parenting Stress Index SF IV | 6 and 12 months after enrollment
  A validated 36 item questionnaire in parents of children older than 1 month assessing child anxiety/mood (Internalizing Symptoms), relationships and attachment and parent, caregiver and family mental health and functioning. Scoring yields an overall stress score and sub-scores for Parental Distress, Parent-Child Dysfunctional Interaction and Difficult Child
Recruitment and Retention Rate | 12 months after enrollment
  Proportion of potential participants who are eligible and enrolled will be tracked. Proportion of individuals with complete data collection at 6 and 12 months will be determined to calculate retention rate.

CONTACTS AND LOCATIONS:
Overall Officials: Imaan Bayoumi, MD, MSc, Principal Investigator — Queen's University
Locations (1):
- Queen's Family Health Team, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to researchers whose proposed use of the data has been approved.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of study results.
Access Criteria: Data will be made available to researchers whose proposed use of the data has been approved.

REFERENCES:
- [Derived] Bayoumi I, Parkin PC, Martin M, Keown-Stoneman CDG, Birken CS, Maguire JL, Borkhoff CM. Connecting Families: Poverty Screening and Financial Support Navigation for Families of Young Children in Primary Care: A Pilot Randomized Controlled Trial. Acad Pediatr. 2025 Jul;25(5):102820. doi: 10.1016/j.acap.2025.102820. Epub 2025 Mar 24. PMID 40139488